CLINICAL TRIAL: NCT06623643
Title: The Investigation of Melatonin and Cortisol Levels in the Saliva of Individuals with Bruxism
Brief Title: "Salivary Melatonin and Cortisol Levels in Individuals with Bruxism"
Status: Not yet recruiting | Type: Observational
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, sema kaya, doctor, Yuzuncu Yil University
Other Study IDs: 2024-10-31
Record Dates: First submitted 2024-10-01; First posted 2024-10-02 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Bruxism
Keywords: melatonin; saliva; cortizol
MeSH Terms: conditions — Bruxism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — The melatonin and cortisol levels in the saliva of patients will be examined. Since saliva will be collected, it contains DNA. However, it will not be used for research purposes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 1: Evaluation of Melatonin and Cortisol Levels in Individuals with Bruxism
  Interventions: Diagnostic Test: The investigation of melatonin and cortisol levels in the saliva
- 2: Evaluation of Melatonin and Cortisol Levels in Individuals without Bruxism
  Interventions: Diagnostic Test: The investigation of melatonin and cortisol levels in the saliva

INTERVENTIONS:
Diagnostic Test: The investigation of melatonin and cortisol levels in the saliva — In the related study, patient data from individuals who visited the Oral and Maxillofacial Radiology clinic at Van Yüzüncü Yıl University Faculty of Dentistry with complaints of bruxism will be used. The diagnosis of bruxism will be made based on clinical data. Diagnoses will be made by Dr. Sema KAYA using clinical findings such as patient history used for the current diagnosis of bruxism, tooth wear, tooth mobility, pain in the temporomandibular joint (TMJ), headaches, pain in the chewing muscles, hypertrophy, and a feeling of fatigue. Before taking the saliva samples, patients will be asked to rinse their mouths with sterile water, and then they will be asked to spit into sterile plastic containers. After approximately 3 mL of saliva is collected, it will be transferred to appropriate Eppendorf tubes and stored at -80°C. Melatonin and cortisol levels will later be analyzed using the enzyme-linked immunosorbent assay (ELISA) method.

SUMMARY:
The effects of the hormones melatonin and cortisol, which play a highly effective role in regulating the sleep-wake cycle, on teeth grinding will be scientifically evaluated. Based on the research results, more effective methods for treating patients suffering from bruxism may be identified.

ELIGIBILITY:
Inclusion Criteria:

- Individuals without any known hormonal diseases, not using antidepressants or medications that could alter saliva content, without degenerative diseases affecting the salivary glands, without cysts or tumors affecting the temporomandibular region, and not undergoing insomnia treatment will be included in the study

Exclusion Criteria:

* Individuals with systemic diseases that affect or may potentially affect saliva content, or those using medications that cause these effects, will not be included in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ndividuals with and without bruxism
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
levels of melatonin | Baseline assessment at the start of the study, follow-up assessments at 3 months and 6 months, with final data collection at 12 months.
  individuals with bruxism
levels of cortisol | Baseline assessment at the start of the study, follow-up assessments at 3 months and 6 months, with final data collection at 12 months.
  individuals with bruxism